CLINICAL TRIAL: NCT05745701
Title: A PHASE 1, OPEN-LABEL, FIXED-SEQUENCE STUDY TO EVALUATE THE EFFECT OF ITRACONAZOLE AND CYCLOSPORINE ON THE SINGLE-DOSE PHARMACOKINETICS OF PF-07081532 IN OVERWEIGHT OR OBESE ADULT PARTICIPANTS
Brief Title: A Drug-Drug Interaction Study to Examine the Impact of Itraconazole and Cyclosporine on PF-07081532 Pharmacokinetics in Overweight or Obese Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C3991041
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-05

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Period 1: PF-07081532 (Active Comparator): Participants will receive PF-07081532 as a single dose on Day 1.
  Interventions: Drug: PF-07081532
- Period 2: Cyclosporine + PF-07081532 (Experimental): Participants will receive a single dose of PF-07081532 and a single dose of cyclosporine on Day 1.
  Interventions: Drug: PF-07081532; Device: Cyclosporine
- Period 3: Itraconazole + PF-07081532 (Experimental): Participants will receive itraconazole daily for 9 days plus a single dose of PF-07081532 on Day 4.
  Interventions: Drug: PF-07081532; Drug: Itraconazole

INTERVENTIONS:
Drug: PF-07081532 — Oral Tablet
Device: Cyclosporine — Oral Solution
  Arms: Period 2: Cyclosporine + PF-07081532
Drug: Itraconazole — Oral Capsule
  Arms: Period 3: Itraconazole + PF-07081532

SUMMARY:
This is a Phase 1, open-label, fixed-sequence, 3-period study to evaluate the effect of multiple doses of itraconazole and a single dose of cyclosporine on the single-dose PK of PF-07081532 in otherwise healthy, overweight or obese, adult female and male participants.

The 3 study periods will be conducted consecutively without a break.

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise healthy female and male participants must be at least 18 years of age at the time of signing the ICD (healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, physical examination, including blood pressure and pulse rate measurement, standard 12-lead ECG and clinical laboratory tests).
2. BMI: ≥25.0 kg/m2 at Screening.
3. Stable body weight, defined as <5 kg change (per participant report) for 90 days before Screening.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Diagnosis of type 1 or type 2 diabetes mellitus or secondary forms of diabetes at Screening.
3. Any malignancy not considered cured (except basal cell carcinoma and squamous cell carcinoma of the skin)
4. Personal or family history of MTC or MEN2, or study participants with suspected MTC per the investigator's judgment.
5. Acute pancreatitis, a history of repeated episodes of acute pancreatitis, or history of chronic pancreatitis.
6. Symptomatic gallbladder disease.
7. Medical history or characteristics suggestive of genetic or syndromic obesity or obesity induced by other endocrinological disorders (eg, Cushing Syndrome).
8. History of depressive disorder or history of other severe psychiatric disorders (eg, schizophrenia or bipolar disorder) within the last 2 years from screening.
9. Known medical history of active liver disease, including chronic hepatitis B or C, primary biliary cirrhosis, alcoholic liver disease, primary sclerosing cholangitis, autoimmune hepatitis, overlap syndrome, or prior known drug-induced liver injury.
10. History of HIV infection.
11. Any lifetime history of a suicide attempt.
12. Use of prohibited medications
13. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest.
14. Standard 12-lead ECG that demonstrates clinically relevant abnormalities that mayaffect participant safety or interpretation of study result.
15. Participants with clinical laboratory test abnormalities at Screening. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3991041

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 16 participants were enrolled in the study. All enrolled participants received 3-period treatments in a fixed sequence. All enrolled participants were treated and completed the study.
Groups:
- Lotiglipron (PF-07081532) Then Lotiglipron + Cyclosporine Then Lotiglipron + Itraconazole: Period 1 (Study Days -1 to 5): Participants received 40 milligram (mg) single dose (SD) lotiglipron orally on Day 1 of Period 1. Period 1 was followed by Period 2.
  Period 2 (Study Days 6 to 10): Participants received 40 mg SD lotiglipron orally and a 600 mg SD cyclosporine orally on Day 1 of Period 2. Period 2 was followed by Period 3.
  Period 3 (Study Days 11 to 20): Participants received 200 mg SD itraconazole orally for 9 days and 40 mg SD lotiglipron orally on Day 4 of Period 3.
  Participants were followed up to maximum of 35 days from the last dose of study intervention.
Period: Period 1: PF-07081532
Arm/Group | Lotiglipron (PF-07081532) Then Lotiglipron + Cyclosporine Then Lotiglipron + Itraconazole
Started | 16
Completed | 16
Not Completed | 0
Period: Period 2: Cyclosporine + PF-07081532
Arm/Group | Lotiglipron (PF-07081532) Then Lotiglipron + Cyclosporine Then Lotiglipron + Itraconazole
Started | 16
Completed | 16
Not Completed | 0
Period: Period 3: Itraconazole + PF-07081532
Arm/Group | Lotiglipron (PF-07081532) Then Lotiglipron + Cyclosporine Then Lotiglipron + Itraconazole
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This group includes all participants who enrolled in this study and received at least 1 dose of study intervention.
Groups:
- Lotiglipron Then Lotiglipron + Cyclosporine Then Lotiglipron + Itraconazole: Period 1 (Study Days -1 to 5): Participants received 40 mg SD lotiglipron orally on Day 1 of Period 1. Period 1 was followed by Period 2.
  Period 2 (Study Days 6 to 10): Participants received 40 mg SD lotiglipron orally and a 600 mg SD cyclosporine orally on Day 1 of Period 2. Period 2 was followed by Period 3.
  Period 3 (Study Days 11 to 20): Participants received 200 mg SD itraconazole orally for 9 days and 40 mg SD lotiglipron orally on Day 4 of Period 3.
  Participants were followed up to maximum of 35 days from the last dose of study intervention.
Arm/Group | Lotiglipron Then Lotiglipron + Cyclosporine Then Lotiglipron + Itraconazole
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.2 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 5
  More than one race | 2
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] — Body Mass Index (kg/m^2) = weight (kg) / [0.01✕height (cm)]^2
  kg/m^2 | 28.6 [25.4 to 37.8]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of Lotiglipron When Administered Alone and With Itraconazole or Cyclosporine
Description: AUCinf is area under the plasma concentration-time profile from time zero extrapolated to infinite time. AUCinf is caluculated by AUClast + (Clast/kel), where Clast is the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis.
Time Frame: Pre-dose of lotiglipron and at 0.5, 1, 2, 4, 6, 8, 10, 12, 14, 24, 36, 48, 72, 96, 120, and 144 (for Period 3 only) hours post dose of lotiglipron on Day 1 of Periods 1 and 2 and on Day 4 of Period 3.
Population: All participants who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of primary interest were reported. The outcome measure was reported by 3 arms to characterize the effect of MD itraconazole and SD cyclosporine on the single dose PK of lotiglipron.
  The 120-hour PK samples collected in Period 1 was the same as the pre-dose PK samples in Periods 2. The 120-hour PK sample from Period 2 was taken on Day 1 of Period 3 prior to itraconazole dose administration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Groups:
- Active Comparator: Period 1: Lotiglipron: Participants received 40 mg SD lotiglipron orally on Day 1 of Period 1.
- Experimental: Period 2: Lotiglipron + Cyclosporine: Participants received 40 mg SD lotiglipron orally and 600 mg SD cyclosporine orally on Day 1 of Period 2.
- Experimental: Period 3: Itraconazole+Lotiglipron: Participants received 200 mg SD itraconazole orally for 9 days plus 40 mg SD lotiglipron orally on Day 4 of Period 3.
Arm/Group | Active Comparator: Period 1: Lotiglipron | Experimental: Period 2: Lotiglipron + Cyclosporine | Experimental: Period 3: Itraconazole+Lotiglipron
Number analyzed (Participants) | 16 | 16 | 16
nanogram*hour/milliliter (ng*hr/mL) | 81800 (49) | 162800 (62) | 212900 (36)
Statistical Analysis 1: Comparison: Active Comparator: Period 1: Lotiglipron vs Experimental: Period 2: Lotiglipron + Cyclosporine; Natural loge transformed Cmax of PF-07081532 administered without cyclosporine (Reference) or coadministered with cyclosporine (Test) were analyzed using a mixed effect model with treatment as a fixed effect and participant as a random effect. Estimates of the adjusted mean differences (Test/Reference) and corresponding 90% CIs was obtained from the models. The ratios (and 90% CIs) were expressed as percentages; Test type: Other; test/reference ratios = 195.90, 90% CI 2-sided [162.13 to 236.71]
Statistical Analysis 2: Comparison: Active Comparator: Period 1: Lotiglipron vs Experimental: Period 3: Itraconazole+Lotiglipron; Natural loge transformed Cmax of PF-07081532 administered without itraconazole (Reference) or coadministered with itraconazole (Test) were analyzed using a mixed effect model with treatment as a fixed effect and participant as a random effect. Estimates of the adjusted mean differences (Test/Reference) and corresponding 90% CIs was obtained from the models. The ratios (and 90% CIs) were expressed as percentages; Test type: Other; test/reference ratios = 282.13, 90% CI 2-sided [258.81 to 307.55]

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious adverse event (SAE) was defined as an AE: 1. resulting in death, 2. was life-threatening, 3. required inpatient hospitalization or prolongation of existing hospitalization, 4. resulted in persistent disability, 5. was a congenital anomaly/birth defect, or considered to be an important medical event. Any AEs occurring following start of treatment were considered as treatment emergent adverse event (TEAE). Events that occur during follow-up within the lag time of up to 35 days after the last dose of study intervention were counted as treatment emergent and attributed to the last treatment taken.
Time Frame: From the first dose up to 35 days after administration of the final dose of study intervention (Period 3 Day 9, Study Day 19), the maximum duration was 54 Days
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Lotiglipron Then Lotiglipron + Cyclosporine Then Lotiglipron + Itraconazole
Number analyzed (Participants) | 16
Participants
  All causality TEAEs | 11
  Treatment-Related TEAEs | 11
  All causality Treatment-emergent SAEs | 0

3. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Participants with laboratory abnormalities (without regard to baseline abnormality) that met pre-specified criteria: For HEMATOLOGY, 1) Erythrocyte (Ery.) Mean Corpuscular Volume (fL) < 0.9*Lower limit of normal (LLN), 2) Ery. Mean Corpuscular Hemoglobin (picograms [pg]/cell) < 0.9*LLN; 3） Eosinophils/Leukocytes (%)> 1.2*upper limit of normal (ULN); for CLINICAL CHEMISTRY, Urate (mg/dL)> 1.2*ULN; for URINALYSIS, Urine Hemoglobin (Scalar)≥ 1.
Time Frame: Baseline (pre-dose on Day 1), Period 2 Day 5 (Study Day 10), and Period 3 Day 10 (Study Day 20)
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Lotiglipron Then Lotiglipron + Cyclosporine Then Lotiglipron + Itraconazole
Number analyzed (Participants) | 16
Participants
  HEMATOLOGY- Ery. Mean Corpuscular Volume (fL) < 0.9*LLN | 1
  HEMATOLOGY-Ery. Mean Corpuscular Hemoglobin (pg/cell) < 0.9*LLN | 1
  HEMATOLOGY-Eosinophils/Leukocytes (%)> 1.2*ULN | 1
  CLINICAL CHEMISTRY-Urate (mg/dL)> 1.2*ULN | 1
  URINALYSIS-URINE Hemoglobin (Scalar)≥ 1 | 1

4. Secondary Outcome: Number of Participants Meeting Pre-Specified Criteria of Vital Signs
Description: Pre-specified criteria of vital signs included: Supine diastolic blood pressure (BP) <50mmHg, change from baseline maximum (max) decrease or increase >=20mmHg; supine pulse rate min< 40 beats per minute (bpm), max> 120 bpm; Supine systolic BP: Value <90 mmHg, change from baseline max decrease or increase >=30mmHg
Time Frame: Pre-dose Day 1 in periods 1, 2 and 3 (Study Days 1, 6, and 11, respectively), and prior to discharge on Period 3 Day 10 (Study Day 20)
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Lotiglipron Then Lotiglipron + Cyclosporine Then Lotiglipron + Itraconazole
Number analyzed (Participants) | 16
Participants | 0

5. Secondary Outcome: Change From Baseline in Body Weight at the End of Periods 1, 2, and 3
Description: Observed value at baseline and change from baseline in body weight at Day 5 of Period 1 , Day 5 of Period 2, and Day 10 of Period 3 were summarized.
Time Frame: Baseline (pre-dose on Day 1), Day 5 of Period 1 (Study Day 5), Day 5 of Period 2 (Study Day 10), and Day 10 of Period 3 (Study Day 20)
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Lotiglipron Then Lotiglipron + Cyclosporine Then Lotiglipron + Itraconazole
Number analyzed (Participants) | 16
Kilogram (kg)
  Baseline | 87.631 (12.9350)
  Day 5 of Period 1 | -1.631 (1.1904)
  Day 5 of Period 2 | -1.956 (1.4778)
  Day 10 of Period 3 | -2.256 (1.6541)

6. Secondary Outcome: Number of Participants Meeting Pre-Specified Criteria of Electrocardiogram (ECGs)
Description: The pre-specified criteria of ECG included: QT interval, aggregated: value >500 millisecond (msec); corrected QT Fridericia method (QTCF) interval, aggregated: 450<=value<480 msec, 480<=value<500 msec, value>=500 msec, 30<=changes<60msec, and changes>=60msec.
Time Frame: as for outcome 4
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Lotiglipron Then Lotiglipron + Cyclosporine Then Lotiglipron + Itraconazole
Number analyzed (Participants) | 16
Participants | 0

7. Secondary Outcome: Number of Participants With Suicidal Ideation or Behavior According to Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is an interview-based rating scale to systematically assess suicidal ideation and suicidal behavior. Participants who respond "yes" to any question related to suicidal ideation or behavioral are reported in this outcome measure.
Time Frame: Period 1 Day -1 (Study Day -1), Period 3 Day 10 (Study Day 20) or Early Termination visit
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Lotiglipron Then Lotiglipron + Cyclosporine Then Lotiglipron + Itraconazole
Number analyzed (Participants) | 16
Participants | 0

8. Secondary Outcome: Number of Participants With a Score of ≥15 on Patient Health Questionnaire-9 (PHQ-9)
Description: PHQ9-9 is a 9 item self-report scale for the assessment of depressive symptoms. A PHQ-9 score of ≥15 indicates clinically significant depression and was reported in this outcome measure. The total score ranges from 0 to 27 with the following interpretation: Score 1-4: minimal depression; Score 5-9: Mild depression; Score 10-14: moderate depression; Score 15-19 moderately severe depression; Score 20-27: Severe depression
Time Frame: Period 1 Day -1 (Study Day -1), Period 3 Day 10 (Study Day 20) or Early Termination visit
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Lotiglipron Then Lotiglipron + Cyclosporine Then Lotiglipron + Itraconazole
Number analyzed (Participants) | 16
Participants | 0

9. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Lotiglipron When Administered Alone and With Itraconazole or Cyclosporine
Description: Cmax is the maximum observed concentration and is observed directly from data.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Active Comparator: Period 1: Lotiglipron | Experimental: Period 2: Lotiglipron + Cyclosporine | Experimental: Period 3: Itraconazole+Lotiglipron
Number analyzed (Participants) | 16 | 16 | 16
nanogram/milliliter (ng/mL) | 4165 (28) | 5207 (35) | 5180 (24)

10. Secondary Outcome: Time to Cmax (Tmax) of Lotiglipron When Administered Alone and With Itraconazole or Cyclosporine
Description: Tmax is the Time to Cmax and is observed directly from data as time of first occurrence.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Groups:
- Active Comparator: Period 1: Lotiglipron: Participants received 40 mg SD lotiglipron orally on Period 1 Day 1.
Arm/Group | Active Comparator: Period 1: Lotiglipron | Experimental: Period 2: Lotiglipron + Cyclosporine | Experimental: Period 3: Itraconazole+Lotiglipron
Number analyzed (Participants) | 16 | 16 | 16
hr | 6.00 [3.98 to 8.00] | 6.00 [2.00 to 12.0] | 5.03 [2.00 to 10.0]

11. Secondary Outcome: Apparent Oral Clearance (CL/F) of Lotiglipron When Administered Alone and With Itraconazole or Cyclosporine
Description: CL/F is the apparent oral clearance and is calculated by Dose/AUCinf.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre (L)/hr
Arm/Group | Active Comparator: Period 1: Lotiglipron | Experimental: Period 2: Lotiglipron + Cyclosporine | Experimental: Period 3: Itraconazole+Lotiglipron
Number analyzed (Participants) | 16 | 16 | 16
Litre (L)/hr | 0.4890 (49) | 0.2458 (62) | 0.1879 (36)

12. Secondary Outcome: Apparent Oral Volume of Distribution (Vz/F) of Lotiglipron When Administered Alone and With Itraconazole or Cyclosporine
Description: Vz/F is the apparent volume of distribution and is calculated by Dose/ (AUCinf*kel), where kel is the terminal phase rate constant calculated by a linear regression of the log linear concentration time curve
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre
Arm/Group | Active Comparator: Period 1: Lotiglipron | Experimental: Period 2: Lotiglipron + Cyclosporine | Experimental: Period 3: Itraconazole+Lotiglipron
Number analyzed (Participants) | 16 | 16 | 16
Litre | 15.01 (31) | 8.261 (47) | 11.91 (28)

13. Secondary Outcome: Terminal Half-life (t1/2) of Lotiglipron When Administered Alone and With Itraconazole or Cyclosporine
Description: T1/2 is calculated by Loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log linear concentration time curve. Only those data points judged to describe the terminal log linear decline were used in the regression.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Active Comparator: Period 1: Lotiglipron | Experimental: Period 2: Lotiglipron + Cyclosporine | Experimental: Period 3: Itraconazole+Lotiglipron
Number analyzed (Participants) | 16 | 16 | 16
hr | 21.96 (6.1239) | 24.14 (7.3865) | 45.02 (9.7607)

ADVERSE EVENTS:
Time Frame: From the first dose up to 35 days after administration of the final dose of study intervention (Period 3 Day 9, Study Day 19), the maximum duration was 54 Days
Arm/Group | Lotiglipron Then Lotiglipron + Cyclosporine Then Lotiglipron + Itraconazole
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 11/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lotiglipron Then Lotiglipron + Cyclosporine Then Lotiglipron + Itraconazole (N=16)
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 4
Eructation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 2
Feeling hot (General disorders) | 6
Scratch (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 4
Dizziness (Nervous system disorders) | 1
Dizziness postural (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Hypoaesthesia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Somatic symptom disorder (Psychiatric disorders) | 1
Chromaturia (Renal and urinary disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Hot flush (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/01/NCT05745701/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT05745701/SAP_001.pdf